CLINICAL TRIAL: NCT06542536
Title: Investigation of Tolerability, Safety, and Pharmacokinetic Properties of a Single Oral Dose of Monlunabant in Male Japanese and Caucasian Participants With Normal Body Weight
Brief Title: A Research Study Investigating Safety and Concentration in the Blood After One Dose Tablet of the New Medicine Monlunabant in Healthy Weight Japanese and Caucasian Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9440-7952; U1111-1299-1093 (Other: World Health Organization (WHO))
Record Dates: First submitted 2024-08-05; First posted 2024-08-07 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Monlunabant dose 1 (Experimental): Dose 1 of monlunabant treatment
  Interventions: Drug: Monlunabant
- Monlunabant dose 2 (Experimental): Dose 2 of monlunabant treatment
  Interventions: Drug: Monlunabant
- Monlunabant dose 3 (Experimental): Dose 3 of the monlunabant treatment
  Interventions: Drug: Monlunabant
- Placebo (monlunabant) (Placebo Comparator): Placebo treatment
  Interventions: Drug: Placebo (monlunabant)

INTERVENTIONS:
Drug: Monlunabant — Oral monlunabant
  Arms: Monlunabant dose 1; Monlunabant dose 2; Monlunabant dose 3
Drug: Placebo (monlunabant) — Oral placebo (monlunabant)
  Arms: Placebo (monlunabant)

SUMMARY:
The study is testing a new study drug in healthy normal weight Japanese and Caucasian participants after a single dose. The aim of this study is to see if the new medicine is safe and how it works in the participants body. Oral monlunabant is a new medicine which cannot be prescribed by doctors but has previously been tested in humans. The participant will either get monlunabant or placebo or a combination of both. Which treatment the participant get is decided by chance. The study will last for about 49 days in total.

ELIGIBILITY:
Inclusion Criteria:

* Male.
* Age 18-55 years (both inclusive) at the time of signing the informed consent.
* Considered eligible based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator.
* For Japanese participants, both parents of Japanese descent and both paternal and maternal grandparents of Japanese descent.
* For Caucasian participants, self-reported European descent or white Latin-American descent.
* BMI 18.5-24.9 kg/m^2 (both inclusive) at screening.

Exclusion Criteria:

* Known or suspected hypersensitivity to study intervention(s) or related products.
* Previous randomisation in this study.
* Previous rescreening for this study.
* History of Major Depressive Disorder within the last 2 years from screening.
* Presence or history of any psychiatric disorders (e.g., schizophrenia, bipolar disorder, eating disorders, depression, and anxiety) as judged by the investigator.
* Suicidal ideation corresponding to type 4 or 5 or suicidal behaviour on the Columbia-Suicide Severity Rating Scale (C-SSRS) as assessed at screening or any history of suicidal attempts.
* A Patient Health Questionnaire 9 (PHQ-9) score greater than 9 as assessed at screening.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2024-08-09 (Actual); Primary Completion 2024-10-25 (Actual); Study Completion 2024-10-25 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events (TEAEs) after single dose of oral monlunabant | From dosing (day 1) to end of study visit (day 21)
  Number of events

SECONDARY OUTCOMES:
AUC0-∞,monlunabant, SD; the area under the monlunabant plasma concentration-time curve from time 0 to infinity after single dose of oral monlunabant | From pre-dose (day 1) to end of study visit (day 21)
  h*nmol/L
Cmax, monlunabant, SD; the maximum plasma concentration of monlunabant after single dose of oral monlunabant | From pre-dose (day 1) to end of study visit (day 21)
  nmol/L
tmax,monlunabant, SD; the time of maximum observed plasma concentration of monlunabant single dose of oral monlunabant | From pre-dose (day 1) to end of study visit (day 21)
  h (hours)
t½,monlunabant,SD; the terminal half-life of monlunabant after single dose of oral monlunabant | From pre-dose (day 1) to end of study visit (day 21)
  h (hours)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Altasciences Clinical LA, Inc., Cypress, California, United States

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com